CLINICAL TRIAL: NCT03281122
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986224 in Healthy Subjects and Chronic Heart Failure Patients With Reduced Ejection Fraction
Brief Title: A Study of BMS-986224 in Healthy Subjects and Heart Failure Patients With Reduced Ejection Fraction
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CV016-007
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): Specified dose on specified days
  Interventions: Drug: Placebo; Drug: BMS-986224
- Arm B (Placebo Comparator): Specified dose on specified days
  Interventions: Drug: Placebo; Drug: BMS-986224

INTERVENTIONS:
Drug: Placebo — Specified dose on specified days
Drug: BMS-986224 — Specified dose on specified days

SUMMARY:
The purpose of this study is test the safety and tolerability of BMS-986224 and its effects on the body in healthy subjects and subjects with chronic heart failure with reduced ejection fraction

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

Healthy Subjects (Part A and B)

* Healthy subjects, as determined by no clinically significant deviations in medical history, physical examination, ECGs, vital signs, and clinical laboratory determinations
* Subjects must be willing and able to complete all study-specific procedures and visits
* Additional criterion for Japanese subjects in Groups BJ1 to BJ3: Subjects must be first generation Japanese (born in Japan and not living outside of Japan for > 10 years, and both parents are ethnically Japanese)

Heart Failure Patients (Part C)

* Left ventricular EF <45% and >25%, as assessed by cardiac MRI within 3 months of first dose of study drug; or left ventricular EF <40% and >25% as assessed by echocardiogram at Screening or within 3 months of first dose of study drug; left ventricular EF
* Heart failure is considered to be stable at the discretion of the Investigator (i.e., no acute cardiovascular [CV] events or hospitalization (including emergency room visits) for CV causes within 3 months of first dose of study drug
* Regular sinus rhythm at Screening and no history of atrial fibrillation in the past 12 months

Exclusion Criteria:

Healthy Subjects (Part A and B)

* Major surgery within 4 weeks of (first) study treatment administration
* Inability to be venipunctured and/or tolerate venous access
* Subjects who have smoked or used smoking cessation or nicotine containing products (including, but not limited, to e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum, varenicline, bupropion) within 6 months of the first dose of study drug

Heart Failure Patients (Part C)

* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption
* Major surgery within 4 weeks of (first) study treatment administration
* Inability to be venipunctured and/or tolerate venous access

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 199 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | Up to one month
Number of Adverse Events (AEs) | Up to one month
Number of deaths | Up to one month

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to one month
Time of maximum observed plasma concentration (Tmax) | Up to one month
Terminal elimination half-life (T-HALF) | Up to one month
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] | Up to one month
Area under the plasma concentration-time curve from time zero extrapoloated [AUC(INF)] | Up to one month
Area under the concentration-time curve in one dosing interval [AUC(TAU)] | Up to one month
Accumulation ratio: ratio of Cmax following last dose to Cmax following first dose (ARcmax) | Up to one month
Accumulation ratio: ratio of AUC(TAU) following last dose to AUC(TAU) following first dose (ARtau) | Up to one month
Terminal elimination rate constant (kel) | Up to one month
Apparent oral clearance, calculated as dose/AUC(INF) for single dose or dose/AUC(TAU) for multiple dose | Up to one month
Apparent volume of distribution at terminal phase (Vz/F) | Up to one month
Cumulative urinary excretion (of the unchanged drug) over one dosing interval [Ae(TAU)] | Up to one month
Cumulative urinary excretion (of the unchanged drug) [Aet] | Up to one month
Renal clearance (CLr) | Up to one month
Amount excreted unchanged (%) [UR%] | Up to one month
Ratio of Metabolite Cmax to Parent Cmax, corrected for molecular weight (MR_Cmax) | Up to one month
Ratio of Metabolite AUC(INF) to Parent AUC(INF), corrected for molecular weight | Up to one month
Ratio of Metabolite AUC(0-T) to Parent AUC(0-T), corrected for molecular weight [MR_AUC(0-T)] | Up to one month
Ratio of Metabolite AUC(TAU) to Parent AUC(TAU), corrected for molecular weight [MR_AUC(TAU)] | Up to one month
Drug-drug interaction (DDI) assessment | Up to one month

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- Czechia (2):
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Krajska zdravotni - Masarykova nemocnice v Usti nad Labem, Ústí nad Labem
- Netherlands (5):
  - Deventer Ziekenhuis, Deventer
  - Universitair Medisch Centrum Groningen, Groningen
  - PRA Health Sciences - Groningen, Groningen
  - Spaarne Gasthuis - Haarlem-Zuid, Haarlem
  - D & A Research and Genetics, Sneek
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny Number 4 w Lublinie, Lublin
  - 4th Wojskowy Szpital Kliniczny z Poliklinika Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Wroclaw
- Spain (5):
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Alvaro Cunqueiro, Vigo
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Tayside, Dundee
  - The University of Edinburgh, Edinburgh
  - Richmond Pharmacology, London

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm